CLINICAL TRIAL: NCT01389245
Title: An Open, Prospective, Multi-center Study to Evaluate the OsseoSpeed™ TX Implant With an Early Loading Protocol in Patients With Tooth Loss in the Posterior Maxilla. A 3-years Follow-up Study.
Brief Title: Study on OsseoSpeed™ TX Implants in the Upper Jaw in a Chinese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-0001
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Partially Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous, Partially

ARMS (1):
- OsseoSpeed™ TX (Experimental): OsseoSpeed™ TX implants of lengths 8-17 mm
  Interventions: Device: OsseoSpeed™ TX

INTERVENTIONS:
Device: OsseoSpeed™ TX — OsseoSpeed™ TX implants of lengths 8-17 mm

SUMMARY:
The purpose of this study is to investigate the clinical efficacy of OsseoSpeed™ TX implants in a Chinese population by evaluation of marginal bone level alteration, implant stability and implant survival in the posterior maxilla up to 3 years after loading. Hypothesis: Early loading of the posterior maxilla is a safe and predictable procedure.

ELIGIBILITY:
Inclusion criteria:

1. Provision of informed consent
2. Aged 20-75 years at enrollment
3. History of edentulism in the posterior maxilla, Kennedy classes I or II, of at least four months. Last natural tooth in function is canine or first bicuspid.
4. Neighboring tooth to the planned bridge must have natural root.
5. Presence of natural teeth, partial prosthesis and/or implants in the opposite jaw in contact with the planned bridge.
6. Deemed by the investigator to have adequate bone height and a bone width of minimum 5.5 mm.
7. Deemed by the investigator as likely to present an initially stable implant situation

Exclusion criteria:

1. Unlikely to be able to comply with study procedures, as judged by the investigator
2. Earlier graft procedures in the study area
3. Current need for pre-surgical bone or soft tissue augmentation in the planned implant area.
4. Uncontrolled pathologic processes in the oral cavity
5. Known or suspected current malignancy
6. History of radiation therapy in the head and neck region
7. History of chemotherapy within 5 years prior to surgery
8. Systemic or local disease or condition that could compromise post-operative healing and/or osseointegration
9. Uncontrolled diabetes mellitus
10. Corticosteroids or any other medication that could influence post-operative healing and/or osseointegration
11. Smoking more than 10 cigarettes/day
12. Present alcohol and/or drug abuse
13. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
14. Previous enrollment in the present study.
15. Simultaneous participation in another clinical study or participation in a clinical study during the last 6 months.
16. Subjects that are unable to give informed consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2015-07 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deng Feilong, MD, Principal Investigator — Guanghua School of Stomatology, Sun Yat-Sen University, Guangzhou
Locations (3):
- China (3):
  - Capital Medical University School of Stomatology, Centre of Oral Implantation, Beijing
  - Guanghua School of Stomatology, Sun Yat-Sen University, Guangzhou
  - Department of Prosthodontics, Nanjing Stomatology Hospital, Nanjing University, Nanjing

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Period: Overall Study
Arm/Group | OsseoSpeed™ TX
Started | 42; 110 Implants
Completed | 27; 66 Implants
Not Completed | 15; 44 Implants
Not completed — Protocol Violation | 10
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population = Per Protocol Population. I.e. Protocol deviators excluded, a total of 10 subjects with 24 implants.
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 32
Number analyzed (Implants) | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18
Region of Enrollment [Count of Participants; unit: Participants]
  China | 32

OUTCOME MEASURES:

1. Primary Outcome: Marginal Bone Level Alteration
Description: Marginal bone level determined from radiographs and expressed as the distance from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal bone level expressed in millimeters at the 3-year follow-up visit compared to values obtained at delivery of permanent restoration i.e. loading (baseline).
Time Frame: Measured at implant loading and at the 3-year follow-up after implant loading.
Population: 36 subjects (86 implants) completed the 3-year follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 27 subjects (66 implants). Eighteen of the radiographs were not possible to evaluate, giving an overall number of 19 subjects (48 implants) as basis for the 3-year Marginal Bone Level alteration analysis.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 19
Number analyzed (Implants) | 48
Millimeter | -0.09 (0.83)

2. Secondary Outcome: Number of Stable Implants
Description: Implant stability evaluated clinically/manually (recorded as stable yes/no).
Time Frame: Measured at the 3-year follow-up after implant loading.
Population: 36 subjects (86 implants) completed the 3-year follow-up visit. Analysis of implant stability was performed on the all patients treated population.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 36
Number analyzed (Implants) | 86
Implants | 86

3. Secondary Outcome: Evaluation of the Periimplant Mucosa Condition - By Assessment of PPD
Description: Condition of the periimplant mucosa by assessment of probing pocket depth (PPD).
  Change in pocket depth expressed in millimeters at the 3-year follow-up visit, compared to values obtained at delivery of permanent restoration, i.e. loading (baseline).
  Negative value = increased pocket depth.
Time Frame: Measured at the 3-year follow-up after implant loading.
Population: 36 subjects (86 implants) completed the 3-year follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 27 subjects (66 implants). For two of those implants evaluation of PPD was not performed, giving 25 subjects (64 implants) as basis for the PPD analysis.
Measure: Mean (Standard Deviation); unit: Millimeter
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 25
Number analyzed (Implants) | 64
Millimeter | -0.23 (0.90)

4. Secondary Outcome: Number of Survived Implants
Description: Implant survival rate evaluated by clinically and radiographically, counting the number of implants remaining in function.
Time Frame: Measured at the 3-year follow-up after implant loading.
Population: All participants treated with at least one study implant.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 42
Number analyzed (Implants) | 110
Implants | 103

5. Secondary Outcome: Presence of Plaque
Description: Occurence of plaque around the study implant. Presented as number of implants that show presence of plaque at time of the 3-year follow-up visit after implant loading.
Time Frame: Measured at the 3-year follow-up after implant loading.
Population: 36 subjects (86 implants) completed the 3-year follow-up visit. Protocol deviations were excluded, giving a per-protocol analysis population of 27 subjects (66 implants). Evaluation of plaque was not performed on two of those subjects, giving an overall number of 25 subjects (64 implants) as basis for the 3-year presence of plaque analysis.
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | OsseoSpeed™ TX
Number analyzed (Participants) | 25
Number analyzed (Implants) | 64
Implants | 9

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | OsseoSpeed™ TX
Serious Adverse Events (participants affected / at risk) | 3/42
Other Adverse Events (participants affected / at risk) | 7/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed™ TX (N=42)
Paralytic stroke (Vascular disorders) | 1 (1)
Adenocarcinoma of urinary bladder (Renal and urinary disorders) | 1 (1)
Femur Neck Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OsseoSpeed™ TX (N=42)
Insufficient osseointegration of the implant during healing phase (Musculoskeletal and connective tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less